CLINICAL TRIAL: NCT02052544
Title: Clinical Performance Evaluation of Pefakit® PiCT® UC In Vitro Diagnostic Medical Device
Status: Completed | Type: Observational
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PICT-01
Record Dates: First submitted 2014-01-17; First posted 2014-02-03 (Estimated); Results first posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Thromboembolic Events
Keywords: determination of heparin levels; Patients; requiring; unfractionated
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study patients: Patients receiving unfractionated heparin (UFH)

SUMMARY:
To demonstrate the substantial equivalence (SE) of Pefakit® PiCT® UC (test device, T) to aPTT-SP (Hemosil) (predicate device, P) in determining heparin levels in subjects undergoing heparin therapy in support of a United States Food and Drug Administration (FDA) 510(k) submission.

DETAILED DESCRIPTION:
Standard of Care Study. Objective is to monitor the patients' heparin levels under treatment with continuous unfractionated heparin infusions. Blood samples collections (4 ml) are required routinely. A proportion of this standard sample (leftover plasma) will be used for study purposes. About three samples will be analyzed which are collected within 2 - 4 days. Time points for blood sample collections will be defined by the treating physician according the local standard of care and will be associated exclusively to clinical considerations. Results of the Pefakit® PiCT® UC assay will NOT be used to take therapeutic decisions for study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects receiving a continuous infusion with UFH
* Subjects who have given written informed consent (unless written informed consent is waived by local regulations or local EC/IRB)

Exclusion Criteria:

* Subjects treated with any other anticoagulants other than UFH
* Subjects who have been undergoing fibrinolytic therapy within the previous 4 weeks
* Subjects who are known to have a congenital bleeding disorder
* Subjects known to present unexplained prolongations of clotting time
* Subjects known to have coagulation factor deficiencies
* Patient participating or who has participated within one month from enrolment in another investigational study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects undergoing UFH anticoagulation therapy will are needed for this study. Typically, such patients are undergoing cardiovascular surgery, are being treated for thromboembolic events, or are receiving heparin intravenously for thrombosis prophylaxis due to its more advantageous pharmacokinetic profile in some situations.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Korte, Principal Investigator — Deputy Head Institute for Clinical Chemistry and Hematology; Manuela K. Krause, MD, Principal Investigator — Deutsche Klinik für Diagnostik GmbH; Rathbun Suman, MD, Principal Investigator — University of Oklahoma Health Sciences Center- Department of Medicine
Locations (3):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States
- Deutsche Klinik für Diagnostik, Wiesbaden, Hesse, Germany
- Cantonal Hospital -Institue for Clinical Chemistry and hematology, Sankt Gallen, Switzerland, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: FPI: Jul 2012; LPO May 2013
  All three centers were hospitals (medical clinics) with certified laboratory.
Pre-assignment Details: Plasma from subjects treated with any other anticoagulants other than UFH. Plasma from subjects who have been undergoing fibrinolytic therapy within the previous 4 weeks.
Period: Overall Study
Arm/Group | Study Patients
Started | 123 (First Subject In)
Completed | 123 (Last Subject Out)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 144 subjects signed ICF. 4 out of 144 failed in/exclusion criteria 123 subjets are part of the AVS (all valid subjects) population. All 123 UFH treated study subjects had previous and concomitant medications and treatments.
Groups:
- Plasma Samples From Subjects Receiving Unfractionated Heparin: A total of 123 valid patients were recruited over three clinical centers (two in Europe, one in the US). The patients were selected from subjects receiving UFH therapy and who have given written informed consent. Excluded from the study were subjects treated with any other anticoagulants other than UFH, subjects who have been undergoing fibrinolytic therapy within the previous 4 weeks, subjects known to have a congenital bleeding disorder, subjects known to show coagulation factor deficiencies and subjects known to have a coagulation inhibitor or an unexplained APTT prolongation.
Arm/Group | Plasma Samples From Subjects Receiving Unfractionated Heparin
Number analyzed (Participants) | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 67
Age, Continuous [Mean (Full Range); unit: years] | 65.5 [18 to 100]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 68
Race/Ethnicity, Customized [Number; unit: partecipants]
  Oriental | 1
  African American | 6
  Caucasian | 114
  Hispanic | 2
Region of Enrollment [Number; unit: participants]
  United States | 51
  Germany | 38
  Switzerland | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Sensitivity and Specificity of Pefakit and Hemosil.
Description: Sensitivity is the proportion of positive cases identified as positive. Specificity is the proportion of negative cases identified as negative. The Sensitivity and Specificity of Pefakit and Hemosil were calculated for the overall study population and separately for each of the three medical centers. Sensitivity and Specificity of Pefakit and Hemosil were each assessed relative to the reference method (Biophen)
Time Frame: within 2 - 4 days
Population: AVS (all valid subjects) population: All valid subjects with no major deviation affecting outcome.413 samples total analyzed
Measure: Number (95% Confidence Interval); unit: percentage of cases
Groups:
- Pefakit: Sensitivity and Specificity of Pefakit
- Hemosil: Sensitivity and Specificity of Hemosil
Arm/Group | Pefakit | Hemosil
Number analyzed (Participants) | 121 | 121
percentage of cases
  Overall Sensitivity% | 83.3 [75.7 to 89.4] | 77 [68.6 to 84]
  Overall Specificity% | 81.5 [68.6 to 90.7] | 59.3 [45 to 72.4]
  site #1 (St.Gallen) Sensitivity% | 90.6 [79.3 to 96.9] | 94.3 [84.3 to 98.8]
  site #1 (St.Gallen) Specificity | 72.7 [39 to 94] | 27.3 [6 to 61]
  site #2 (Wiesbaden) Sensitivity% | 74.4 [58.8 to 86.5] | 53.5 [37.7 to 68.8]
  site #2 (Wiesbaden) Specificity% | 78.3 [56.3 to 92.5] | 69.6 [47.1 to 86.8]
  site #3 (Oklahoma) Sensitivity% | 83.3 [65.3 to 94.4] | 80 [61.4 to 92.3]
  site #3 (Oklahoma) Specificity% | 90 [68.3 to 98.8] | 65 [40.8 to 84.6]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of FPI (first patient in) until LPO (last patient out).
Description: In the US the study meets the requirements for exemption as defined in the Investigational Device Exemption regulations (21 CFR Part 812.2(c)).
  In the EU, national regulations were followed regarding adverse event reporting for IVD studies.
Arm/Group | Study Patients
Serious Adverse Events (participants affected / at risk) | 0/123
Other Adverse Events (participants affected / at risk) | 0/123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any proposed publication, lecture, manuscript, poster presentation or other disclosure or dissemination of the data or Results of this study by PI shall be submitted to DSM at least forty-five (45) days prior to its submission for publication or use for DSM's review, comment and approval. DSM reserves the right to have deleted from the proposed text all of DSM's Confidential Information which may be contained therein. DSM's comments shall be provided without undue delay.